CLINICAL TRIAL: NCT05937477
Title: Developing Artificial Intelligence-based Algorism Based on Life-log Data Acquired From Wearable Device for the Prediction of Chemotherapy-induced Side Effects and Symptom
Brief Title: Developing Artificial Intelligence-based Algorism to Predict Side Effects and Symptoms From Chemotherapy
Status: Recruiting | Type: Observational
Sponsor: Sehhoon Park (Other)
Responsible Party: Sponsor-Investigator, Sehhoon Park, M.D, Ph.D. Principal Investigator, Clinical Professor, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Other Study IDs: 2023-02-057
Record Dates: First submitted 2023-06-14; First posted 2023-07-10 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Lung Cancer; Head and Neck Cancer; Esophageal Cancer
MeSH Terms: conditions — Lung Neoplasms; Head and Neck Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neoadjuvant, Adjuvant Chemotherapy Arm: Patients diagnosed with lung, head and neck, or esophageal cancer and undergoing Neoadjuvant, Adjuvant chemotherapy.
  Interventions: Other: Fitbit smartwatch
- Palliative Chemotherapy Arm: Patients diagnosed with lung, head and neck, or esophageal cancer and undergoing Palliative chemotherapy.
  Interventions: Other: Fitbit smartwatch

INTERVENTIONS:
Other: Fitbit smartwatch — Patients wear the wearable to check their biomarkers and use the application to assess their quality of life and side effects at one-week intervals.

SUMMARY:
In this study, the investigators obtain wearable disease based biomarkers from patients diagnosed with cancer and undergoing chemotherapy, and simultaneously measure patient self-reported adverse events through an app to evaluate chemotherapy completion rates, emergency room visits, and frequency of CTCAE adverse events.

The investigators will develop an artificial intelligence-based algorism that can predict patients' side effects based on biomarkers alone.

DETAILED DESCRIPTION:
In this study, patients diagnosed with lung, head and neck, and esophageal cancers and undergoing chemotherapy will be measured for self-reported side effects using a wearable device to collect biomarkers through an app, and the association between patient quality of life and side effects and biomarkers obtained from the wearable device will be analyzed. On the other hand, blood (EDTA 3cc) for pharmacogenomics testing will be tested once at any point during the study period as an indicator associated with side effects after chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 20 years of age or older
* Must have diagnosed with lung, head and neck, or esophageal cancer,

  1. scheduled to receive their first treatment in preoperative or postoperative chemotherapy.
  2. scheduled for systemic chemotherapy due to recurrence or metastasis.
* Eastern Cooperative Oncology (ECOG) performance status of 0 to 2.
* Patients who have access to a smartphone and can use the mobile app on their own.
* Understand the purpose of the study and agree to participate in the study.

Exclusion Criteria:

* Patients who, in the judgment of the researcher, have difficulty using the application.
* Patients who are judged by the medical staff to be unable to participate in the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing chemotherapy after being diagnosed with lung, head and neck, or esophageal cancer.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-06-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Developing artificial intelligence prediction algorism | Through study completion, an average of 30 months
  PRO data and treatment information collected from the wearable are used to evaluate correlations through methods such as linear regression to determine valid variables, utilizing LSTM models, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Gangnamgu, South Korea